CLINICAL TRIAL: NCT01513551
Title: A Multicenter, Double-Blind Study of the Safety, Tolerability, and Immunogenicity of a Pneumococcal Conjugate Vaccine (V114) Compared to Pneumococcal Polysaccharide Vaccine (PNEUMOVAX® 23) and PREVNAR 13® (Pneumococcal 13-Valent Conjugate Vaccine [Diphtheria CRM197 Protein]) in Healthy Adults 50 Years of Age or Older
Brief Title: The Safety, Tolerability, and Immunogenicity Profiles of a Single Dose of V114, PNEUMOVAX® 23, or PREVNAR 13® in Adults 50 Years of Age or Older (V114-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-002; 2011-004542-18 (Other: EudraCT Number); V114-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-12-27; First posted 2012-01-20 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal vaccines
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- V114 (Experimental): Healthy adult participants received a single 0.5 mL intramuscular injection of aluminum adjuvanted V114 on Day 1.
  Interventions: Biological: Pneumococcal Conjugate Vaccine (V114)
- PNEUMOVAX® 23 (Active Comparator): Healthy adult participants received a single 0.5 mL intramuscular injection of PNEUMOVAX® 23 on Day 1.
  Interventions: Biological: PNEUMOVAX® 23
- PREVNAR 13® (Active Comparator): Healthy adult participants received a single 0.5 mL intramuscular injection of PREVNAR 13® on Day 1.
  Interventions: Biological: PREVNAR 13®

INTERVENTIONS:
Biological: Pneumococcal Conjugate Vaccine (V114) — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and aluminum phosphate adjuvant (125 mcg) in each 0.5 mL dose.
  Arms: V114
Biological: PNEUMOVAX® 23 — 23-valent pneumococcal polysaccharide vaccine with serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F (25 mcg each) in each 0.5 mL dose.
  Arms: PNEUMOVAX® 23
Biological: PREVNAR 13® — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F, serotype 6B (4.4 mcg each) and aluminum phosphate adjuvant (125 mcg) in each 0.5. mL dose.
  Arms: PREVNAR 13®

SUMMARY:
The purpose of the study is to see if an investigational vaccine for Streptococcus pneumonia disease (V114) has comparable safety, tolerability, and antibody response to Pneumococcal Polysaccharide Vaccine (PNEUMOVAX® 23) and 13-valent Pneumococcal Conjugate Vaccine (PREVNAR 13®) when administered to healthy adults 50 years of age or older.

The primary hypothesis is the serotype-specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) as measured by the pneumococcal electrochemiluminescence (Pn ECL) assay at one month postvaccination in subjects who receive V114 will be noninferior to those measured in subjects who receive PNEUMOVAX® 23.

ELIGIBILITY:
Inclusion Criteria:

-Without fever for 72 hours prior to vaccination

Exclusion Criteria:

* Prior receipt of any pneumococcal polysaccharide vaccine or any pneumococcal conjugate vaccine
* Known or suspected to be immunocompromised
* Functional or anatomic asplenia
* History of autoimmune disease
* Evidence of dementia or cognitive impairment
* Use of any immunosuppressive therapy
* Received a licensed non-live vaccine administered within the 14 days prior to receipt of study vaccine or scheduled to receive any other licensed vaccine within 30 days following receipt of study vaccine
* Received a licensed live virus vaccine within 30 days prior of receipt of study vaccine or is scheduled to receive any other licensed vaccine within 30 days of receipt of study vaccine
* Received any vaccine containing diphtheria toxoid within 6 months prior to receipt of study vaccine
* Received a blood transfusion or blood products within the 6 months before receipt of study vaccine or scheduled to receive a blood transfusion or blood product within 30 days of receipt of study vaccine
* History of invasive pneumococcal disease or known history of other culture-positive pneumococcal disease
* Received antibiotic therapy for any acute illness within 72 hours before receipt of study vaccine

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2013-02-15 (Actual); Study Completion 2013-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ermlich SJ, Andrews CP, Folkerth S, Rupp R, Greenberg D, McFetridge RD, Hartzel J, Marchese RD, Stek JE, Abeygunawardana C, Musey LK. Safety and immunogenicity of 15-valent pneumococcal conjugate vaccine in pneumococcal vaccine-naive adults >/=50 years of age. Vaccine. 2018 Oct 29;36(45):6875-6882. doi: 10.1016/j.vaccine.2018.03.012. Epub 2018 Mar 17. PMID 29559167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 25 trial centers: 10 in the United States; 2 in Canada; 2 in Denmark; 2 in Israel; 2 in Norway, 3 in Poland, 2 in Spain and 2 in Sweden.
Period: Overall Study
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Started | 230 | 231 | 231
Vaccinated | 230 | 231 | 230
Completed | 226 | 225 | 226
Not Completed | 4 | 6 | 5
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 5 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Randomized but not vaccinated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all randomized participants who received study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13® | Total
Number analyzed (Participants) | 230 | 231 | 230 | 691
Age, Customized [Count of Participants; unit: Participants]
  50 to 64 years | 79 | 80 | 80 | 239
  65 to 74 years | 75 | 76 | 74 | 225
  >= 75 years | 76 | 75 | 76 | 227
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 123 | 122 | 367
  Male | 108 | 108 | 108 | 324
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 20 | 14 | 48
  Not Hispanic or Latino | 216 | 211 | 215 | 642
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 5 | 6 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 10 | 6 | 12 | 28
  White | 212 | 217 | 212 | 641
  More than one race | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the Sponsor's product, is also an adverse experience.
Time Frame: All AEs: up to 14 days after vaccination; Serious Adverse Events (SAEs): up to 6 months after vaccination
Population: The analysis population consisted of those participants who received study vaccination and had safety follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 229 | 230 | 230
Percentage of Participants | 75.1 | 68.3 | 65.7
Statistical Analysis 1: Comparison: V114 vs PNEUMOVAX® 23; Test type: Other; Miettinen & Nurminen; Risk Difference (RD) = 6.8, 95% CI 2-sided [-1.4 to 15.0]
Statistical Analysis 2: Comparison: V114 vs PREVNAR 13®; Test type: Other; Miettinen & Nurminen; Risk Difference (RD) = 9.5, 95% CI 2-sided [1.1 to 17.7]

2. Primary Outcome: Percentage of Participants With an Injection-site Adverse Event Reported With >=2% Incidence in One or More Vaccination Groups
Description: Injection-site AEs reported by >=2% of participants in one or more vaccination groups were assessed.
Time Frame: Up to Day 14 postvaccination
Population: The analysis population consisted of those participants who received study vaccination and had safety follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 229 | 230 | 230
Percentage of Participants
  Injection site erythema | 14.8 | 14.8 | 13.0
  Injection site induration | 14.8 | 10.4 | 12.6
  Injection site pain | 60.3 | 51.3 | 53.0
  Injection site pruritus | 3.1 | 1.3 | 2.2
  Injection site swelling | 20.1 | 10.9 | 18.3
  Injection site warmth | 0.9 | 0.0 | 2.2

3. Primary Outcome: Percentage of Participants With a Systemic Adverse Event Reported With >=2% Incidence in One or More Vaccination Groups
Description: Systemic AEs reported by >=2% of participants in one or more vaccination groups were assessed.
Time Frame: Up to Day 14 postvaccination
Population: The analysis population consisted of those participants who received study vaccination and had safety follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 229 | 230 | 230
Percentage of Participants | 48.5 | 43.9 | 45.6

4. Primary Outcome: Percentage of Participants With a Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to 6 months postvaccination
Population: The analysis population consisted of those participants who received study vaccination and had safety follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 229 | 230 | 230
Percentage of Participants | 1.7 | 3.0 | 2.2

5. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A SAE is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. SAEs deemed by the investigator to be possibly, probably, or definitely related to study vaccine were reported.
Time Frame: Up to 6 months postvaccination
Population: The analysis population consisted of those participants who received study vaccination and had safety follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 229 | 230 | 230
Percentage of Participants | 0.0 | 0.0 | 0.0

6. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG) Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence (ECL) assay.
Time Frame: One month postvaccination
Population: The analysis population consisted of those participants who were not considered to have violated important protocol requirements that could have impacted the validity of the antibody response measured following vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 210 | 207 | 212
µg/mL
  Serotype 1 | 3.76 [3.05 to 4.65] | 3.30 [2.68 to 4.07] | 3.12 [2.54 to 3.82]
  Serotype 3 | 1.13 [0.96 to 1.35] | 0.57 [0.47 to 0.68] | 0.56 [0.47 to 0.66]
  Serotype 4 | 1.96 [1.59 to 2.41] | 1.03 [0.83 to 1.27] | 2.09 [1.70 to 2.56]
  Serotype 5 | 3.99 [3.23 to 4.92] | 2.70 [2.21 to 3.30] | 2.76 [2.21 to 3.44]
  Serotype 6A: number analyzed (Participants) | 209 | 207 | 212
  Serotype 6A | 4.88 [3.73 to 6.39] | 1.14 [0.90 to 1.43] | 4.86 [3.86 to 6.13]
  Serotype 6B | 5.43 [4.11 to 7.17] | 2.01 [1.58 to 2.57] | 2.81 [2.19 to 3.62]
  Serotype 7F | 4.59 [3.72 to 5.66] | 3.74 [3.00 to 4.65] | 6.06 [4.91 to 7.48]
  Serotype 9V | 4.05 [3.32 to 4.93] | 2.72 [2.21 to 3.36] | 3.41 [2.77 to 4.20]
  Serotype 14 | 8.56 [6.86 to 10.69] | 8.13 [6.38 to 10.36] | 8.90 [7.08 to 11.18]
  Serotype 18C | 8.00 [6.62 to 9.68] | 4.66 [3.73 to 5.82] | 6.83 [5.68 to 8.20]
  Serotype 19A | 9.36 [7.66 to 11.44] | 6.99 [5.67 to 8.61] | 11.36 [9.28 to 13.92]
  Serotype 19F | 3.35 [2.67 to 4.21] | 4.17 [3.32 to 5.24] | 4.80 [3.81 to 6.04]
  Serotype 22F | 5.21 [4.25 to 6.39] | 1.98 [1.61 to 2.44] | 0.38 [0.32 to 0.44]
  Serotype 23F | 5.55 [4.33 to 7.12] | 1.82 [1.44 to 2.30] | 3.41 [2.62 to 4.43]
  Serotype 33F | 11.56 [9.27 to 14.40] | 8.26 [6.52 to 10.47] | 0.85 [0.70 to 1.03]

7. Secondary Outcome: Geometric Mean Titer (GMT) of Pneumococcal Serotype-specific Opsonophagocytic Activity (OPA) Antibodies
Description: OPA for the serotypes contained in V114 was determined using a Multiplex Opsonophagocytic Assay (MOPA-4)
Time Frame: One month postvaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
Number analyzed (Participants) | 210 | 207 | 212
Titer
  Serotype 1: number analyzed (Participants) | 210 | 207 | 211
  Serotype 1 | 208.03 [156.36 to 276.78] | 117.87 [87.11 to 159.49] | 115.75 [85.72 to 156.31]
  Serotype 3: number analyzed (Participants) | 210 | 207 | 210
  Serotype 3 | 595.16 [498.23 to 710.95] | 313.83 [256.64 to 383.76] | 256.76 [212.08 to 310.85]
  Serotype 4: number analyzed (Participants) | 209 | 206 | 211
  Serotype 4 | 2875.79 [2215.61 to 3732.69] | 1099.88 [804.01 to 1504.63] | 3001.63 [2380.57 to 3784.72]
  Serotype 5: number analyzed (Participants) | 210 | 207 | 211
  Serotype 5 | 712.21 [537.78 to 943.22] | 288.41 [210.03 to 396.06] | 372.35 [271.76 to 510.19]
  Serotype 6A: number analyzed (Participants) | 207 | 201 | 211
  Serotype 6A | 4216.34 [2977.07 to 5971.49] | 490.60 [325.94 to 738.44] | 5251.47 [4114.87 to 6702.00]
  Serotype 6B: number analyzed (Participants) | 209 | 206 | 210
  Serotype 6B | 6469.99 [4775.27 to 8766.16] | 1630.20 [1174.34 to 2263.03] | 4207.86 [3212.46 to 5511.70]
  Serotype 7F: number analyzed (Participants) | 210 | 206 | 209
  Serotype 7F | 5148.66 [4170.62 to 6356.06] | 3665.62 [2722.58 to 4935.30] | 7816.74 [6358.89 to 9608.81]
  Serotype 9V: number analyzed (Participants) | 208 | 205 | 208
  Serotype 9V | 3024.34 [2338.72 to 3910.96] | 1674.44 [1252.72 to 2238.12] | 2471.10 [1882.58 to 3243.60]
  Serotype 14: number analyzed (Participants) | 210 | 207 | 209
  Serotype 14 | 4352.27 [3374.62 to 5613.15] | 3572.27 [2667.12 to 4784.61] | 4478.38 [3647.04 to 5499.22]
  Serotype 18C: number analyzed (Participants) | 209 | 205 | 211
  Serotype 18C | 4631.86 [3730.53 to 5750.96] | 2438.57 [1839.33 to 3233.04] | 3358.41 [2665.75 to 4231.06]
  Serotype 19A: number analyzed (Participants) | 210 | 206 | 211
  Serotype 19A | 3391.18 [2755.18 to 4174.00] | 2682.65 [2095.62 to 3434.12] | 4186.28 [3421.20 to 5122.46]
  Serotype 19F: number analyzed (Participants) | 208 | 206 | 209
  Serotype 19F | 1201.17 [906.20 to 1592.15] | 1581.60 [1211.55 to 2064.67] | 1946.04 [1547.41 to 2447.35]
  Serotype 22F: number analyzed (Participants) | 208 | 203 | 197
  Serotype 22F | 8329.52 [6542.87 to 10604.06] | 4382.78 [3359.60 to 5717.58] | 57.45 [37.29 to 88.50]
  Serotype 23F: number analyzed (Participants) | 208 | 206 | 210
  Serotype 23F | 2217.18 [1588.99 to 3093.71] | 378.41 [262.42 to 545.67] | 1197.80 [836.80 to 1714.53]
  Serotype 33F: number analyzed (Participants) | 210 | 207 | 210
  Serotype 33F | 31116.90 [24612.69 to 39339.94] | 27560.15 [21471.19 to 35375.88] | 3129.94 [2441.58 to 4012.38]

ADVERSE EVENTS:
Time Frame: Up to 6 months postvaccination
Description: The at-risk population consisted of all participants who received study vaccination and had safety follow-up.
Arm/Group | V114 | PNEUMOVAX® 23 | PREVNAR 13®
All-Cause Mortality (participants affected / at risk) | 0/229 | 1/230 | 0/230
Serious Adverse Events (participants affected / at risk) | 4/229 | 7/230 | 5/230
Other Adverse Events (participants affected / at risk) | 167/229 | 149/230 | 141/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=229) | PNEUMOVAX® 23 (N=230) | PREVNAR 13® (N=230)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=229) | PNEUMOVAX® 23 (N=230) | PREVNAR 13® (N=230)
Fatigue (General disorders) | 57 (68) | 63 (89) | 55 (75)
Injection site erythema (General disorders) | 34 (37) | 34 (34) | 30 (31)
Injection site induration (General disorders) | 34 (35) | 24 (24) | 29 (29)
Injection site pain (General disorders) | 138 (145) | 118 (126) | 122 (137)
Injection site swelling (General disorders) | 46 (48) | 25 (26) | 42 (42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (45) | 26 (37) | 29 (41)
Myalgia (Musculoskeletal and connective tissue disorders) | 69 (74) | 60 (72) | 50 (60)
Headache (Nervous system disorders) | 40 (43) | 41 (55) | 42 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.